CLINICAL TRIAL: NCT00508638
Title: Improving Heart Failure Risk Stratification in the ED
Brief Title: Identifying High- and Low-Risk Heart Failure Patients in the Emergency Department (The Stratify Study)
Acronym: Stratify
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Cincinnati (Other)
Responsible Party: Principal Investigator, Alan Storrow, Vice Chairman for Research and Academic Affairs, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 508; R01HL088459 (NIH); R01 HL055459
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases
Keywords: Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
People with heart failure (HF) symptoms who are seen in the emergency department (ED) are often admitted to the hospital even though it may not be necessary. This study will gather information from HF patients seen in the ED to develop a decision-making tool that will help doctors predict the risk of HF-related death or serious complications. Improving the ability of ED doctors to effectively and safely manage low-risk HF patients should lead to fewer unnecessary hospitalizations.

DETAILED DESCRIPTION:
HF is a life-threatening condition in which the heart can no longer pump enough blood to the rest of the body. Symptoms of HF can include shortness of breath, nausea, fatigue, swelling of the feet or abdomen, and an irregular or rapid pulse. A critical challenge facing ED doctors is how to best manage people who come into the ED with symptoms of HF. Currently, most people evaluated for HF in the ED are admitted to the hospital; however, not all of these people are in need of such intensive treatment. It is estimated that up to 50% of HF-related hospital admissions could be avoided. Improving the ability of the ED doctor to effectively and safely manage low-risk HF patients is essential to avoid unnecessary hospitalizations. This study will gather information from ED patients at risk for HF to develop an algorithm decision tool that will predict patients' risk for inpatient or outpatient death and serious complications from HF. This decision tool will be distributed worldwide for ED use and will hopefully reduce the costs of HF care by appropriately allocating hospital resources.

This study will enroll adults admitted to the ED with possible signs of HF. While in the ED, participants will undergo a digital heart sound recording procedure, a medical record review, blood collection, and a brief cognitive assessment. Five and 30 days following the ED visit, participants will be contacted by phone or will be visited in the hospital by study staff. Information will be collected on health status and unplanned hospital or ED visits that have occurred following the initial ED visit.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the adult ED with difficulty breathing, peripheral edema, or fatigue
* Meets Framingham criteria for congestive heart failure
* Willing and able to give informed consent; this will be determined based on participants' ability to remain in a conscious state, ability to remain awake, ability to ask questions about the study or answer questions that are asked, and ability to date and sign a consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a convenience sample of patients presenting to the emergency department for care.
Sampling Method: Non-Probability Sample
Enrollment: 1033 (Actual)
Dates: Start 2007-05; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Information collected from participants while in the hospital, including a digital heart sound recording procedure, a medical record review, blood collection, and a brief cognitive assessment | Measured while participants are in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Alan B. Storrow, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Collins SP, Hart KW, Lindsell CJ, Fermann GJ, Weintraub NL, Miller KF, Roll SN, Sperling MI, Sawyer DB, Storrow AB. Elevated urinary neutrophil gelatinase-associated lipocalcin after acute heart failure treatment is associated with worsening renal function and adverse events. Eur J Heart Fail. 2012 Sep;14(9):1020-9. doi: 10.1093/eurjhf/hfs087. Epub 2012 Jun 25. PMID 22733980
- [Background] Collins SP, Lindsell CJ, Storrow AB, Fermann GJ, Levy PD, Pang PS, Weintraub N, Frank Peacock W, Sawyer DB, Gheorghiade M. Early changes in clinical characteristics after emergency department therapy for acute heart failure syndromes: identifying patients who do not respond to standard therapy. Heart Fail Rev. 2012 May;17(3):387-94. doi: 10.1007/s10741-011-9294-7. PMID 22160814
- [Background] Pang PS, Collins SP, Storrow AB. Letter by Pang et al regarding article, "Early deaths in heart failure patients discharged from the emergency department: a population-based analysis". Circ Heart Fail. 2010 Jul;3(4):e22; author reply e23. doi: 10.1161/CIRCHEARTFAILURE.110.945865. No abstract available. PMID 20647481
- [Result] Collins SP, Lindsell CJ, Yealy DM, Maron DJ, Naftilan AJ, McPherson JA, Storrow AB. A comparison of criterion standard methods to diagnose acute heart failure. Congest Heart Fail. 2012 Sep-Oct;18(5):262-71. doi: 10.1111/j.1751-7133.2012.00288.x. Epub 2012 Apr 4. PMID 22994440
- [Derived] Doering A, Jenkins CA, Storrow AB, Lindenfeld J, Fermann GJ, Miller KF, Sperling M, Collins SP. Markers of diuretic resistance in emergency department patients with acute heart failure. Int J Emerg Med. 2017 Dec;10(1):17. doi: 10.1186/s12245-017-0143-x. Epub 2017 May 8. PMID 28484958
- [Derived] Collins SP, Jenkins CA, Harrell FE Jr, Liu D, Miller KF, Lindsell CJ, Naftilan AJ, McPherson JA, Maron DJ, Sawyer DB, Weintraub NL, Fermann GJ, Roll SK, Sperling M, Storrow AB. Identification of Emergency Department Patients With Acute Heart Failure at Low Risk for 30-Day Adverse Events: The STRATIFY Decision Tool. JACC Heart Fail. 2015 Oct;3(10):737-47. doi: 10.1016/j.jchf.2015.05.007. PMID 26449993
- [Derived] Collins SP, Lindsell CJ, Jenkins CA, Harrell FE, Fermann GJ, Miller KF, Roll SN, Sperling MI, Maron DJ, Naftilan AJ, McPherson JA, Weintraub NL, Sawyer DB, Storrow AB. Risk stratification in acute heart failure: rationale and design of the STRATIFY and DECIDE studies. Am Heart J. 2012 Dec;164(6):825-34. doi: 10.1016/j.ahj.2012.07.033. Epub 2012 Oct 29. PMID 23194482